CLINICAL TRIAL: NCT02031926
Title: Evaluation of the Reproductibility of the Pressure Generated by a Positive Expiratory Pressure Device
Brief Title: Evaluation of Correct PEP Use With the Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Physiotherapist, PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEP training
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
MeSH Terms: interventions — Positive-Pressure Respiration

ARMS (1):
- Positive expiratory pressure (Experimental)
  Interventions: Device: Positive expiratory pressure

INTERVENTIONS:
Device: Positive expiratory pressure

SUMMARY:
Healthy subjects will be trained to used correctly a positive expiratory pressure device. The aim of the study is to evaluate te reproductibility of the correct used of the device after training

ELIGIBILITY:
Inclusion Criteria:

* No lung disease
* Older than 18 years

Exclusion Criteria:

* Psychological disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Expiratory pressure | within the 7 first days

SECONDARY OUTCOMES:
Succes rate | Every day

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium